CLINICAL TRIAL: NCT06317688
Title: Effectiveness of Highly Purified Anhydrous (HPA) Lanolin Versus Extra-Virgin Coconut Oil in Preventing Subacute Lactation Mastitis
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Harris Health System (Houston, Texas) (Unknown)
Responsible Party: Principal Investigator, Sonia Riley, PhD Candidate, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TWU IRB-FY2023-157
Record Dates: First submitted 2023-11-08; First posted 2024-03-19 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Lactation Mastitis; Breast Feeding; Staphylococcus Aureus Infection
MeSH Terms: conditions — Breast Feeding; Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial- Random Assignment-Random Selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pre-Screening (No Intervention): Pre-Screening to meet qualifications and conditions of study.
- Demographic Data Stage I (No Intervention): Data information gathered for enrollment
- Demographic Data StageII (No Intervention): Data gathered after delivery
- Clinical Data (Experimental): 50%Administration of Extra-Virgin Coconut Oil/ 50% HPA Lanolin
  Interventions: Dietary Supplement: Extra-Virgin Coconut Oil

INTERVENTIONS:
Dietary Supplement: Extra-Virgin Coconut Oil — Active ingredients act as a destructor of bacteria, viruses and fungus
  Other Names: HPA Lanolin (Attention Control)
  Arms: Clinical Data

SUMMARY:
Problem of the Study This study was designed to test the effectiveness of the application of extra-virgin coconut oil versus Highly Purified Anhydrous (HPA) Lanolin in ameliorating nipple pain, cracking and eventually the prevention of subacute lactation mastitis in breastfeeding women. It is theorized that the nipple crack, nipple pain are early warning signs of subacute clinical lactation mastitis. Goal is after application of extra-virgin coconut oil comparative analysis will be done at one week, three weeks, and six weeks. These complications associated with development of subacute mastitis can be addressed early during the first six weeks of lactation.

DETAILED DESCRIPTION:
Lanolin is the standard of care in many healthcare institutions. However, lanolin is not supported by the literature as a gold standard of treatment and care. Frequent dermatoses reactions as well as the lack of wound healing and its use as a protective barrier was not found sufficient to promote effective breastfeeding. The origin of lanolin as an animal by product is not ideal supplement for baby's first exposure to a supplement. Furthermore, there is lack of evidential support that lanolin can in fact promote wound healing.

Several studies have been conducted comparing lanolin to other treatments. A representative selection of these studies is presented here. A 2012 study of 100 breastfeeding women was conducted by Dennis et al., 2012, Lanolin was compared to an All-Purpose Nipple Ointment (combination of Mupirocin Ointment 2%, Betamethasone ointment 0.1%, Miconazole 2%) The researchers hypothesized that the combination of creams would target all the known causes of subacute clinical mastitis including fungal infection, atopic dermatitis reactions, staphylococcus aureus infections. The attention control in the double blinded randomized control trial was HPA purified Lanolin. Participants in both the lanolin group and the all-purpose nipple ointment group experienced severe dermal reactions from the topical application. It was concluded that both products were not effective for preventing complications during lactation but rather contributing to the complication of dermatoses.

Another study conducted by Niazi on a sample of 100 breastfeeding women tested the effects of Purslane cream with an attention control of Lanolin which is current practice and found that lanolin in fact doesn't possess wound healing properties but rather has protective barrier properties that are not necessarily intended for promotion of wound healing. Study participants in the purslane group had rapid repair of the nipple and were able to feed more frequently which maintained adequate milk supply and had a more fulfilling experience. Whereas the Lanolin group experiences less frequent feedings, more pain, and often decreased their duration of breastfeeding.

Jackson conducted a study in Ontario Canada of 186 breastfeeding women using a randomized control design to assess the effects of lanolin on nipple pain. No studies to date had assessed HPA Lanolin effects on nipple pain. Group assignment was randomized. An attention control group received latch education as an intervention while the experimental group used Lanolin on their breasts. Breastfeeding self-efficacy, pain rating and maternal satisfaction with lanolin was measured within the study. Lanolin was found to be no more effective than latch treatment group. The lanolin had short-term protective factors but did not promote wound healing. However, women in the study did report high satisfaction with the ease of use of HPA Lanolin.

Hildebrandt conducted a study of 50 postpartum women where the women were their own control nothing was applied to one nipple and HPA Lanolin was applied to the other. The women were monitored for 10 days postpartum, and they were asked to measure or report their pain twice a day using the nipple tenderness scale. The women in this study reported less nipple pain on the lanolin treated breast than on the breast that received no treatment. Similar to the study published by Jackson et al., (2017) Lanolin has some protective factors for short periods of time. Neither study went beyond 10 days of breastfeeding which makes it difficult to assess the long-term effects over the ideal breastfeeding time period.

Properties of Extra-Virgin Coconut Oil This research study is proposing to introduce a topical source that has within the product naturally the properties needed to prevent the complications not solved by traditional methods. Extra-virgin Coconut oil is feasible alternative solution that will promote wound healing, decrease incidence of dermatoses, and is nutritionally fit for baby. Although extra-virgin coconut oil has not been specifically studied in lactating women it has been studied in other areas that can prove its properties (Abbas et al, 2017). These include antimicrobial, antiviral and antifungal effects as well as anti-inflammatory benefits, and the ability to rebuild collagen.

Theoretical Framework The theoretical framework is based on the Grand Theory of Jean Watson's Caring Science The Philosophy and Science of Nursing. Watson Grand Theory of Caring Science underpins this research study as her theory is foundational to nursing. Watson stated that "The ultimate goal of nursing care, Caring Science, and research are to deliver quality, human care" (p.110). The processes described by the Caring Science Theory are systematic and scientific. They follow logical systematic approaches based upon proven methodologies. To accomplish this, science alone is not enough to attract the consumer and create an environment of caring. 'It takes an integration of all forms of creativity, intuition, aesthetics, ethical, personal and sometimes spiritual processes as well as professional empirical technical processes' (p. 107) Methodology Research Questions The following research question is proposed for this research study. Does the topical application of extra-virgin coconut oil to nipples before and after each breast feeding reduce pain and formation of nipple cracks within the first six weeks of lactation more effectively than the topical application of HPA Lanolin? H1- The topical application of extra-virgin coconut oil to nipples before and after each breastfeeding result in a greater reduction in nipple pain during the first six weeks of lactation when compared to the topical application of HPA Lanolin to the same areas.

H2- The topical application of extra-virgin coconut oil to nipples before and after each breastfeeding result in a greater reduction in nipple cracks during the first six weeks of lactation when compared to the topical application of HPA Lanolin to the same area.

Research Design A randomized control experimental design will be used to collect data. The participants will be randomized by random selection. Participants will be randomized to either the experimental group which will receive EVCO or the control group which will receive standard practice of Lanolin. Randomization will occur by the researcher who will divide each into two equal groups. Qualtrics simple excel sheet for randomization will deploy in the randomization process.

Treatment of Data Statistical tests will be analyzed using the SPSS software system version 23. Data will be extracted from Red Cap application and placed into excel spread sheet for easy upload into the SPSS system. Data will be deidentified when used within the SPSS software system. Demographic information will be measured using basic descriptive statistics. These include frequencies, percentages, means and standard deviations. A priori power analysis was conducted using G*Power 3.1.9 to determine the minimum sample size required to find statistical significance using a 2 (group) x 3 (time) repeated measures analysis of variance (i.e., a mixed-model ANOVA). With a desired level of power set at 0.80, alpha (a) level at .05, and a small to moderate effect size of .15 (f), it was determined that a minimum of 74 total participants would be required to ensure adequate power. To account for a 15 % attrition rate, 100 participants will be recruited to ensure adequate power. The research question will also be addressed using a Mann Whitney U (non-parametric t-test) for repeated measure independent samples which will measure significance between the repeated measures taken at one week, three weeks, and six weeks. Post Hoc parametric will use the mixed-model ANOVA which is a more statically stronger test for internal validity if there is a statistically significant differences between the extra-virgin coconut oil and the lanolin group. The fisher's Least significant Difference (LSD) will be employed for the post hoc analysis.

Hypothesis 1 will be measured operationally by comparing week one, week three, and week six using the Mann Whitney U the non-parametric t-test comparing the pain level during the six weeks.

Hypothesis 2 will measure operationally the nipple crack during the one week, three week and six weeks using the Mann Whitney U nonparametric t-test comparing the Nipple Tenderness Scale of the extra-virgin coconut oil group to the HPA Lanolin group.

Data Collection Data collection will begin during the clinic phase of the recruitment process. Women who are pregnant and within the age of 18-45 will be approached during 38-40 weeks' gestation during their prenatal appointments. Signage will be placed in the lobby on a bulletin board or a free-standing aisle. Participants will be asked to scan the QR code on the flyer and complete the pre-screening process. If a participant is missed at the clinic setting, they can be approached within the acute care setting. They will be required to complete the pre-screening process at that point. Complete informed consent for approval and participation.

Once potential participants meet the inclusion criteria and qualify to be enrolled in the study, they will sign an electronic consent form using the Qualtrics system, be assigned an ID number (1-200) and then complete the demographic data form. At time of discharge the research pharmacist will dispense a six-week supply of Lanolin for the control group or a six-week supply of EVCO for the experimental group and instructed on the use of the product by applying a pea size before and after each feeding. Data will be collected electronically via SMS text message on the NTS/NPS at one week, three weeks, and six weeks of breastfeeding.

During hospital admission, the participant's chart will be labeled with a notification of their enrollment for staff to be aware. The participants who are in the experimental group will not be provided with lanolin during their hospital stay. The physician residents will write order for patient to participate in the research study as either the control or experimental. Each participant will be randomized by primary investigator. (Please see diagram for algo rhythm of distribution in Appendix A).

Conclusions The research study seeks to employ a new and innovative technique to ameliorate nipple pain and the nipple crack during lactation and prevent subacute lactation mastitis. The goal of the research is to employ a new technique that has benefits to mother and baby with immediate results. Research has shown that breastmilk is best for baby during the first six months of life. To ensure that the experience is fulfilling and without disease it is important to minimize the potential of untoward circumstances that prevent a fulfilling experience. By randomization, of the women into two groups or rather randomized control trial design the researcher will be able to identify if the cream will be effective in both preventing nipple pain and reducing the incidence of nipple crack.

ELIGIBILITY:
Inclusion Criteria:

* Given Birth and breastfeeding infant at least 50% of time

Exclusion Criteria:

* Not breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-08-14 (Estimated); Study Completion 2024-08-14 (Estimated)

PRIMARY OUTCOMES:
Measurement of change in pain level (Numeric Pain Rating Scale McCaffery, 1989) | Six weeks
  The application should reduce the amount of pain at site
Measurement of Development of Nipple Crack (Nipple Tenderness Scale Storr 1988) | Six weeks
  Application should or is hypothesized to reduce the incidence of development of a nipple crack

CONTACTS AND LOCATIONS:
Locations (1):
- Harris Health System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] References Abbas, A. A., Assikong, E.B., Akeh, M., Upla, P., Tuluma, T.K. (2017). Antimicrobial activity of coconut oil and its derivative (Lauric Acid) on some selected clinical isolates. International Journal of Medical Science and Clinical Inventions (4)8, 3173-3177. https://Doi:10.18535/ijmsci/v4i8.12.
- [Result] As'adi N, Kariman N, Mojab F, Pourhoseingholi MA. The effect of Saqez (Pistacia atlantica) ointment on nipple fissure improvement in breastfeeding women during one-month follow-up. Avicenna J Phytomed. 2017 Nov-Dec;7(6):477-485. PMID 29299430
- [Result] Barbosa-Cesnik C, Schwartz K, Foxman B. Lactation mastitis. JAMA. 2003 Apr 2;289(13):1609-12. doi: 10.1001/jama.289.13.1609. No abstract available. PMID 12672715
- [Result] Dayrit CS. Coconut Oil in Health and Disease: Its and Monolaurin's Potential as Cure for HIV/AIDS. XXXVII Cocotech Meeting. Chennai, India. July 25, 2000.
- [Result] Hildebrandt, E., & Spangler, A. (1993). The effect of modified lanolin on nipple Pain/Damage during the first ten days of breastfeeding. International Journal of Childbirth Education, 8(3), 15-19. Retrieved from https://search.proquest.com/docview/212864505?accountid=45853.
- [Result] Jackson KT, Dennis CL. Lanolin for the treatment of nipple pain in breastfeeding women: a randomized controlled trial. Matern Child Nutr. 2017 Jul;13(3):e12357. doi: 10.1111/mcn.12357. Epub 2016 Aug 1. PMID 27477840
- [Result] Joshi S, Kaushik V, Gode V, Mhaskar S. Coconut Oil and Immunity: What do we really know about it so far? J Assoc Physicians India. 2020 Jul;68(7):67-72. PMID 32602684
- [Result] Kim S, Jang JE, Kim J, Lee YI, Lee DW, Song SY, Lee JH. Enhanced barrier functions and anti-inflammatory effect of cultured coconut extract on human skin. Food Chem Toxicol. 2017 Aug;106(Pt A):367-375. doi: 10.1016/j.fct.2017.05.060. Epub 2017 May 28. PMID 28564614
- [Result] Lavergne NA. Does application of tea bags to sore nipples while breastfeeding provide effective relief? J Obstet Gynecol Neonatal Nurs. 1997 Jan-Feb;26(1):53-8. doi: 10.1111/j.1552-6909.1997.tb01507.x. PMID 9017547
- [Result] Nevin KG, Rajamohan T. Effect of topical application of virgin coconut oil on skin components and antioxidant status during dermal wound healing in young rats. Skin Pharmacol Physiol. 2010;23(6):290-7. doi: 10.1159/000313516. Epub 2010 Jun 3. PMID 20523108
- [Result] Niazi A, Yousefzadeh S, Rakhshandeh H, Esmaily H, Askari VR. Promising effects of purslane cream on the breast fissure in lactating women: A clinical trial. Complement Ther Med. 2019 Apr;43:300-305. doi: 10.1016/j.ctim.2019.02.002. Epub 2019 Feb 7. PMID 30935548
- [Result] Ogbolu DO, Oni AA, Daini OA, Oloko AP. In vitro antimicrobial properties of coconut oil on Candida species in Ibadan, Nigeria. J Med Food. 2007 Jun;10(2):384-7. doi: 10.1089/jmf.2006.1209. PMID 17651080
- [Result] Verallo-Rowell VM, Dillague KM, Syah-Tjundawan BS. Novel antibacterial and emollient effects of coconut and virgin olive oils in adult atopic dermatitis. Dermatitis. 2008 Nov-Dec;19(6):308-15. PMID 19134433
- [Result] Watson, J. (2008). The Philosophy and Science of Caring. University Press of Colorado.
- [Result] Zarshenas M, Zhao Y, Poorarian S, Binns CW, Scott JA. Incidence and Risk Factors of Mastitis in Shiraz, Iran: Results of a Cohort Study. Breastfeed Med. 2017 Jun;12:290-296. doi: 10.1089/bfm.2016.0153. Epub 2017 Apr 18. PMID 28418698